CLINICAL TRIAL: NCT06615401
Title: Understanding Perceived Access and Receipt of Gender-affirming Treatments Among Transgender Veterans
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IIR 22-201
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Gender Dysphoria
Keywords: transgender; gender dysphoria; gender-affirming treatment
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Transgender and Gender Diverse Veterans: Veterans with documentation of either a gender identity disorder diagnoses, self-identified gender identity as transgender and gender diverse or transgender-related health factor.

SUMMARY:
Transgender Veterans (trans Vets) frequently experience gender dysphoria or distress related to discord between their gender identity and birth sex. Gender-affirming treatments (GATs) are medically necessary treatments to reduce gender dysphoria. However, not much is known about the barriers and facilitators that influence GAT access and receipt in VA and VA Community Care (CC), among trans Vets who desire GATs. The goals of this mixed-methods study are to determine which GATs trans Vets receive and in which setting, identify barriers and facilitators associated with desired GAT receipt in VA and CC, examine association of GAT receipt, specifically mental healthcare and hormone therapy, with mental health and suicide risk and understand trans Vet experiences related to receipt and desire for mental healthcare and hormone therapy in VA and CC.

DETAILED DESCRIPTION:
Background: Transgender people experience discord between their gender identity and birth sex, defined as gender dysphoria. Gender-affirming treatments (GATs) are medically necessary treatments to reduce gender dysphoria. However, among transgender Veterans (trans Vets) who desire GATs, not much is known about barriers and facilitators to accessing and receiving GATs in VA and VA Community Care (CC). To ensure effective and equitable GAT access for trans Vets, it is critical to understand: [1] GATs trans Vets receive and where they receive them, [2] barriers, including social determinants of health (SDOH) barriers that are highly prevalent among trans Vets, and facilitators associated with desired GAT receipt in VA and CC, [3] association of GAT receipt, specifically mental healthcare and hormone therapy with mental health and suicide risk , and [4] experiences related to receipt of mental healthcare and hormone therapy in VA and CC .

Significance: This study addresses the 2022 HSR&D priority areas of Access to Care, Health Equity/SDOH, MISSION Act, and research gap of underserved LGBTQ+ Veterans. It is also a high priority for our operational partners in VA LGBTQ+ Health Program, Pharmacy Benefits Management, Office of Integrated Veteran Care, and Office of Mental Health and Suicide Prevention. Knowledge gained from this study will ensure that GAT delivery in the VA is patient-centered and is responsive to the lived realities and needs of trans Vets.

Innovation and Impact: This study will be the first to characterize the GATs received in VA and/or CC to understand how VA and CC are balanced in terms of delivering GATs. This study will also provide novel data on trans Vet experiences related to GAT access in CC and on services and resources used by trans Vets to address barriers that influence GAT access.

Specific Aims: We propose a sequential explanatory mixed method study whose aims are to:

Aim 1. Characterize the GATs received by trans Vets in VA and/or CC (VA/CC) Aim 2. Identify barriers and facilitators associated with desired GAT receipt in VA and CC Aim 3a: Explore association of mental healthcare and hormone with mental health and suicide risk.

Aim 3b. Understand trans Vet experiences related to mental healthcare and hormone therapy in VA and CC.

Methodology: Database Aim 1: We will expand our VA cohort of 9,608 trans Vets (IIR 17-238) from 2006-18 to the data available at the time of funding. We will add CC data to determine the types of GATs received by trans Vets in VA and/or CC. Survey Aim 2: We will survey a national sample of trans Vets identified from Aim 1. Among trans Vets who desire GATs, we will determine SDOH barriers, other barriers, and facilitators associated with desired GAT receipt. Among trans Vets who did not desire GATs, we will determine reasons for not wanting GATs. Aim 3a: Existing survey data from the Aim 2 and linked survey-VA Corporate Data Warehouse will allow robust examination of associations between clinical factors (e.g. co-morbidities), non-clinical factors (e.g. demographics), mental health outcomes (e.g. depression), and suicide risk (e.g. suicide ideation) based on receipt/non-receipt of treatment (mental healthcare, hormone therapy). Aim 3b. Using Aim 2 survey free text responses, we will construct themes related to the experience of trans Vets for mental healthcare and hormone therapy in VA and CC.

Next Steps/Implementation: The proposed study will provide key insights related to the health of trans Vets, while adhering to the new guidance provided within the Forms, Publications, Guidance and Documents Action Team business rules released in April 2025.

ELIGIBILITY:
Inclusion Criteria:

* All veterans with documentation of gender identity disorder diagnoses
* Self-reported gender identity as transgender and relevant transgender-related health factor

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All transmasculine, transfeminine and non-binary Veterans identified by the inclusion criteria above.
Study Population: Transgender and gender diverse veterans as identified by documentation of gender identity disorder diagnoses, self-identified gender identity and transgender-related health factors.
Sampling Method: Non-Probability Sample
Enrollment: 986 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-18 (Actual); Study Completion 2025-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guneet K. Jasuja, PhD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (1):
- VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jasuja GK, Zocchi MS, Reisman JI, Brady JE, Livingston NA, Blosnich JR, Vimalananda VG, Singh RS, Goodman M, Silverberg MJ, Wormwood JB, Shipherd JC. Using Self-Identified Gender Identity Data to Advance Health Equity Among Transgender and Gender Diverse Veterans in the Veterans Health Administration. Med Care. 2025 Nov 1;63(11):833-841. doi: 10.1097/MLR.0000000000002195. Epub 2025 Sep 26. PMID 41001883

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transgender and Gender Diverse Veterans
Started | 986
Completed | 923
Not Completed | 63

BASELINE CHARACTERISTICS:
Arm/Group | Transgender and Gender Diverse Veterans
Number analyzed (Participants) | 986
Age, Customized [Count of Participants; unit: Participants]
  Categorical Age: Under 30 | 199
  Categorical Age: 30 - 39 | 297
  Categorical Age: 40 - 49 | 158
  Categorical Age: 50 - 59 | 127
  Categorical Age: 60 - 69 | 91
  Categorical Age: 70 and over | 51
  Categorical Age: Missing | 63
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Trans Woman/Trans Feminine/Female | 489
  Gender Identity: Trans Man/Trans Masculine/Male | 164
  Gender Identity: Non-Binary and/or Gender Diverse | 191
  Gender Identity: More than one Gender Identity | 122
  Gender Identity: Missing | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 21
  Race/Ethnicity: Black/African American | 37
  Race/Ethnicity: Hispanic/Latino (Any Race) | 89
  Race/Ethnicity: White | 667
  Race/Ethnicity: More than one race | 71
  Race/Ethnicity: Other | 25
  Race/Ethnicity: Missing | 76

OUTCOME MEASURES:

1. Primary Outcome: Receipt of Gender Affirming Treatment
Description: Through a national survey, the investigators will identify receipt of gender-affirming treatment in VA and VA Community Care among transgender and gender diverse Veterans.
Time Frame: About 3.5 months
Population: Receipt of different Gender Affirming Therapy (GAT) is reported only among the population of Veterans who wanted that specific GAT.
Measure: Count of Participants; unit: Participants
Arm/Group | Transgender and Gender Diverse Veterans
Number analyzed (Participants) | 986
Participants
  Received Hormone Therapy: number analyzed (Participants) | 909
  Received Hormone Therapy | 769
  Received Mental Health Care: number analyzed (Participants) | 827
  Received Mental Health Care | 687
  Received Hair Removal: number analyzed (Participants) | 687
  Received Hair Removal | 292
  Received Prosthetics: number analyzed (Participants) | 638
  Received Prosthetics | 468
  Received Vocal Therapy: number analyzed (Participants) | 698
  Received Vocal Therapy | 350
  Received Pre-op Visits: number analyzed (Participants) | 751
  Received Pre-op Visits | 224
  Received Top Surgery: number analyzed (Participants) | 695
  Received Top Surgery | 153
  Received Bottom Surgery: number analyzed (Participants) | 595
  Received Bottom Surgery | 77
  Received Facial Therapy: number analyzed (Participants) | 585
  Received Facial Therapy | 37
  Received Trachea Therapy: number analyzed (Participants) | 361
  Received Trachea Therapy | 29
  Received Post-op Visits: number analyzed (Participants) | 629
  Received Post-op Visits | 127

ADVERSE EVENTS:
Time Frame: About 3.5 months
Arm/Group | Transgender and Gender Diverse Veterans
All-Cause Mortality (participants affected / at risk) | 2/986
Serious Adverse Events (participants affected / at risk) | 0/986
Other Adverse Events (participants affected / at risk) | 0/986

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT06615401/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT06615401/ICF_000.pdf